CLINICAL TRIAL: NCT03588091
Title: A Randomized, Muticenter Double-blind Phase III Study of Neoadjuvant Pyrotinib Plus Trastuzumab and Docetaxel Compared With Placebo Plus Trastuzumab and Docetaxel in Women With HER2 Positive Early Stage or Locally Advanced Breast Cancer
Brief Title: Neoadjuvant Study of Pyrotinib in Combination With Trastuzumab in Patients With HER2 Positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-BLTN-III-NeoBC
Record Dates: First submitted 2018-06-18; First posted 2018-07-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pyrotinib; Trastuzumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- arm1 (Experimental): Pyrotinib Plus trastuzumab and docetaxel
  Interventions: Drug: Pyrotinib; Drug: Trastuzumab; Drug: Docetaxel
- arm2 (Placebo Comparator): placebo plus trastuzumab and docetaxel
  Interventions: Drug: Placebo Oral Tablet; Drug: Trastuzumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Pyrotinib — pyrotinib: 400mg orally daily;
  Arms: arm1
Drug: Placebo Oral Tablet — placebo: 400mg orally daily;
  Arms: arm2
Drug: Trastuzumab — trastuzumab:8mg/kg iv load followed by 6mg/kg iv 3-weekly for a total of 4 cycles;
Drug: Docetaxel — docetaxel:after the biological window, 100mg/m2 for a total of 4 cycles

SUMMARY:
This is a randomised, double-blind multicenter Phase III study for evaluating the efficacy and safety of neoadjuvant pyrotinib and trastuzumab plus docetaxel versus placebo and trastuzumab plus docetaxel given as neoadjuvant treatment in HER2 positive early stage or locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* female patients, 18 years ≤ age ≤ 75 years；
* Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1
* Histologically confirmed invasive breast cancer（early stage or locally advanced）:Primary tumour greater than 2 cm diameter
* HER2 positive (HER2+++ by IHC or FISH+)
* Known hormone receptor status.
* Cardiovascular:Baseline left ventricular ejection fraction (LVEF)≥55% measured by ECHO
* Signed informed consent form (ICF)

Exclusion Criteria:

* metastatic disease (Stage IV) or inflammatory breast cancer
* Previous or current history of malignant neoplasms, except for curatively treated:Basal and squamous cell carcinoma of the skin,Carcinoma in situ of the cervix.
* clinically relevant cardiovascular disease:Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension ≥180/110);
* Unable or unwilling to swallow tablets.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Pathological Complete Response (pCR) at the Time of Surgery evaluated by independent review committee(IRC) | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Percentage of Participants With Pathological Complete Response (pCR) at the Time of Surgery evaluated by sites | Approximately 4 months from randomization following surgery or early withdrawal, whichever occurred first (Surgery was performed within 2 weeks after Cycle 4,each cycle is 21 days)
Event-free survival(EFS) | Following surgery until Year 3
Disease-free Survival (DFS) | Following surgery until Year 3
Distance Disease-free Survival (DDFS) | Following surgery until Year 3
Objective Response Rate (ORR) during neoadjuvant period | Baseline up to cycle 4 (assessed at Baseline, at the time of pre-surgery)up to approximately 12 months

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yet-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The affiliated cancer hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan
  - Huai'an First People's Hospital, Huaian, Jiangsu
  - JiangSu Province Hospital, Nanjing, Jiangsu
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital Of Qingdao University, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital Of Xi'an Jiaotong University, Xian, Shanxi
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Wu J, Jiang Z, Liu Z, Yang B, Yang H, Tang J, Wang K, Liu Y, Wang H, Fu P, Zhang S, Liu Q, Wang S, Huang J, Wang C, Wang S, Wang Y, Zhen L, Zhu X, Wu F, Lin X, Zou J. Neoadjuvant pyrotinib, trastuzumab, and docetaxel for HER2-positive breast cancer (PHEDRA): a double-blind, randomized phase 3 trial. BMC Med. 2022 Dec 27;20(1):498. doi: 10.1186/s12916-022-02708-3. PMID 36575513